CLINICAL TRIAL: NCT04065399
Title: A Phase 1/2, Open-label, Dose-Escalation and Dose-Expansion Cohort Study of SNDX-5613 in Patients With Relapsed/Refractory Leukemias, Including Those Harboring an MLL/KMT2A Gene Rearrangement or Nucleophosmin 1 (NPM1) Mutation
Brief Title: A Study of Revumenib in R/R Leukemias Including Those With an MLL/KMT2A Gene Rearrangement or NPM1 Mutation
Acronym: AUGMENT-101
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-5613-0700; 2020-004104-34 (EudraCT Number)
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Mixed Lineage Acute Leukemia; Mixed Phenotype Acute Leukemia; Acute Leukemia of Ambiguous Lineage
Keywords: AML; ALL; MPAL; MLAL; ALAL; relapsed leukemia; refractory leukemia; acute leukemia; KMT2A; NPM1
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia | interventions — revumenib; Cobicistat

STUDY DESIGN:
Intervention Model Description: Phase 1 will employ an accelerated titration design. The dose escalation will follow a modified Fibonacci sequence.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Revumenib (Experimental): Phase 1: Oral revumenib; sequential cohorts of escalating dose levels of revumenib to identify the MTD and RP2D. Participants will be enrolled in 1 of 6 dose-escalation arms:
  * Arm A: Participants not receiving any strong CYP3A4 inhibitor/inducers or fluconazole
  * Arm B: Participants receiving any strong CYP3A4 inhibitors for antifungal prophylaxis
  * Arm C: Participants receiving revumenib and cobicistat
  * Arm D: Participants receiving fluconazole for antifungal prophylaxis
  * Arm E: Participants not receiving any weak, moderate, or strong CYP3A4 inhibitors/inducers
  * Arm F: Participants receiving isavuconazole for antifungal prophylaxis
  Phase 2: Oral revumenib; Following the determination of the RP2D in Phase 1, 3 indication-specific expansion cohorts will be enrolled as follows:
  * Cohort 2A: Participants with KMT2Ar ALL/MPAL
  * Cohort 2B: Participants with KMT2Ar AML
  * Cohort 2C: Participants with NPM1m AML
  Interventions: Drug: revumenib; Drug: cobicistat

INTERVENTIONS:
Drug: revumenib — revumenib orally
  Other Names: SNDX-5613
Drug: cobicistat — Phase 1 Arm C participants will receive 150 mg cobicistat daily.

SUMMARY:
Phase 1 dose escalation will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of revumenib in participants with acute leukemia.

In Phase 2, participants will be enrolled in 3 indication-specific expansion cohorts to determine the efficacy, short- and long-term safety, and tolerability of revumenib.

DETAILED DESCRIPTION:
Phase 1: Oral revumenib; sequential cohorts of escalating dose levels of revumenib to identify the MTD and RP2D. Participants will be enrolled in one of six dose-escalation arms:

Arm A: Participants not receiving any strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducers or fluconazole.

Arm B: Participants receiving itraconazole, ketoconazole, posaconazole, or voriconazole (strong CYP3A4 inhibitors) for antifungal prophylaxis.

Arm C: Participants receiving revumenib and cobicistat.

Arm D: Participants receiving fluconazole (moderate CYP3A4 inhibitor) for antifungal prophylaxis.

Arm E: Participants not receiving any weak, moderate, or strong CYP3A4 inhibitors/inducers.

Arm F: Participants receiving isavuconazole (moderate CYP3A4 inhibitor) for antifungal prophylaxis.

In Phase 2, participants will be enrolled in 3 indication-specific expansion cohorts to determine the efficacy, short- and long-term safety, and tolerability of revumenib:

* Cohort 2A: Participants with KMT2Ar acute lymphoblastic leukemia (ALL)/mixed phenotype acute leukemia (MPAL)
* Cohort 2B: Participants with KMT2A AML
* Cohort 2C: Participants with NPM1m AML

ELIGIBILITY:
Inclusion Criteria:

Participants must have active acute leukemia (bone marrow blasts ≥5% or reappearance of blasts in peripheral blood) as defined by the National Comprehensive Cancer Network (NCCN) in the NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) for Acute Lymphoblastic Leukemia (Version 1.2020) and Acute Myeloid Leukemia (Version 3.2020), or acute leukemia harboring KMT2A rearrangement, NUP98 rearrangement, or NPM1 mutation that have detectable disease in the bone marrow.

1. Phase 1:

   * Arm A: Participants not receiving any strong CYP3A4 inhibitor/inducers or fluconazole.
   * Arm B: Participants receiving itraconazole, ketoconazole, posaconazole, or voriconazole (strong CYP3A4 inhibitors) for antifungal prophylaxis.
   * Arm C: Participants receiving revumenib in combination with cobicistat.
   * Arm D: Participants receiving fluconazole (moderate CYP3A4 inhibitor).
   * Arm E: Participants not receiving any weak, moderate, or strong CYP3A4 inhibitors/inducers.
   * Arm F: Participants receiving isavuconazole (moderate CYP3A4 inhibitor) for antifungal prophylaxis.
2. Phase 2:

   Documented R/R active acute leukemia (bone marrow blasts ≥5% or reappearance of blasts in peripheral blood) as defined by the NCCN Guidelines® for Acute Lymphoblastic Leukemia (Version 1.2020) and Acute Myeloid Leukemia (Version 3.2020).
   * Cohort 2A: Documented R/R ALL/MPAL with KMT2A rearrangement.
   * Cohort 2B: Documented R/R AML with KMT2A rearrangement.
   * Cohort 2C: Documented R/R AML with NPM1m.
3. White blood cell count below 25,000/ microliter at time of enrollment. Participants may receive cytoreduction prior to enrollment per protocol-specified criteria.
4. Male or female participants aged ≥30 days old.
5. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2 or Karnofsky/Lansky score ≥50.
6. Any prior treatment-related toxicities resolved to ≤Grade 1 prior to enrollment, with the exception of ≤Grade 2 neuropathy or alopecia.
7. Radiation Therapy: At least 60 days from prior total body irradiation (TBI), craniospinal radiation and/or ≥50% radiation of the pelvis, or at least 14 days from local palliative radiation therapy (small port).
8. Stem Cell Infusion: At least 60 days must have elapsed from hematopoietic stem cell transplant and at least 4 weeks must have elapsed from donor lymphocyte infusion.
9. Immunotherapy: At least 42 days since prior immunotherapy, including tumor vaccines, and at least 21 days since receipt of chimeric antigen receptor therapy or other modified T or NK cell therapy.
10. Antileukemia Therapy: At least 14 days, or 5 half-lives, whichever is shorter, since the completion of antileukemic therapy.
11. Hematopoietic Growth Factors: At least 7 days since the completion of therapy with short-acting hematopoietic growth factors and 14 days with long-acting growth factors.
12. Biologics: At least 90 days, or 5 half-lives, whichever is shorter, since the completion of therapy with an antineoplastic biologic agent.
13. Steroids: At least 7 days since systemic glucocorticoid therapy, unless receiving physiologic dosing or cytoreductive therapy.
14. Adequate organ function.
15. If of childbearing potential, willing to use a highly effective method of contraception or double barrier method from the time of enrollment through 120 days following the last study drug dose.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for study participation:

1. Diagnosis of active acute promyelocytic leukemia.
2. Isolated extramedullary relapse (Phase 2 only).
3. Active central nervous system disease (cytologic, such as any blasts on cytospin, or radiographic).
4. Detectable human immunodeficiency virus (HIV) viral load within the previous 6 months. Participants with a known history of HIV 1/2 antibodies must have viral load testing prior to study enrollment.
5. Hepatitis B or C.
6. Pregnant or nursing women.
7. Cardiac Disease:

   * Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
   * Corrected QT interval (QTc) >450 milliseconds.
8. Gastrointestinal Disease:

   * any gastrointestinal issue of the upper GI tract that might affect oral drug absorption or ingestion (that is, gastric bypass, gastroparesis, etc).
   * Cirrhosis with a Child-Pugh score of B or C.
9. Graft-Versus-Host Disease (GVHD): Signs or symptoms of acute or chronic GVHD >Grade 0 within 4 weeks of enrollment. All transplant participants must have been off all systemic immunosuppressive therapy and calcineurin inhibitors for at least 4 weeks prior to enrollment. Participants may be on physiological doses of steroids.
10. Concurrent malignancy in the previous 2 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (for example, breast carcinoma, cervical cancer in situ, melanoma in situ) treated with potentially curative therapy, or concurrent low-grade lymphoma, that is asymptomatic and lacks bulky disease and shows no evidence of progression, and for which the participant is not receiving any systemic therapy or radiation.
11. In Phase 1 and Phase 2: Participants requiring the concurrent use of medications known or suspected to prolong the QT/QTc interval, with the exception of drugs with low risk of QT/QTc prolongation that are used as standard supportive therapies (for example, diphenhydramine, famotidine, ondansetron, Bactrim) and the azoles permitted in the relevant arms of Phase 1 and in Phase 2.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (DLTs) (Phase 1) | Approximately 1 year
  Assessed by the NCI CTCAE version 5.0 (Phase 1)
Number of participants with treatment-emergent adverse events (TEAEs) (Phase 1) | Approximately 1 year
  Assessed by the NCI CTCAE version 5.0 (Phase 1)
Cmax (Phase 1) | Approximately 1 year
  Maximum plasma concentration (Cmax) of revumenib and relevant metabolites (Phase 1)
Tmax (Phase 1) | Approximately 1 year
  Time to observed maximum plasma concentration of revumenib and relevant metabolites (Phase 1)
AUC0-t (Phase 1) | Approximately 1 year
  Area under the plasma concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of revumenib and relevant metabolites (Phase 1)
CR+CRh rate (Phase 2) | Approximately 3 years
  To assess the complete remission (CR) and complete remission with partial hematologic recovery (CRh) rate (Phase 2)
Number of participants with TEAEs (Phase 2) | Approximately 3 years
  Assessed by the NCI CTCAE version 5.0 (Phase 2)

SECONDARY OUTCOMES:
Transfusion independence (Phase 2) | Approximately 3 years
  Transfusion independence is defined as any transfusion-free period lasting for at least 56 consecutive days
CRc rate (Phase 2) | Approximately 3 years
  To assess the composite definition of complete remission (CRc) rate (Phase 2)
ORR (CRc+ morphological leukemia-free state [MLFS] + partial remission [PR]) (Phase 2) | Approximately 3 years
  To assess the overall response rate (ORR) of revumenib (Phase 2)
TTR (Phase 2) | Approximately 34 months
  To assess the time to response (TTR) of revumenib (Phase 2)
DOR (Phase 2) | Approximately 3 years
  To assess the duration of response (DOR) of revumenib (Phase 2)
EFS (Phase 2) | Approximately 3 years
  To assess the event free survival (EFS) of revumenib (Phase 2)
OS (Phase 2) | Approximately 5 years
  To assess overall survival (OS) of revumenib (Phase 2)
Cmax (Phase 2) | Approximately 3 years
  Cmax of revumenib and relevant metabolites (Phase 2)
Tmax (Phase 2) | Approximately 3 years
  Tmax of revumenib and relevant metabolites (Phase 2)
AUC0-t (Phase 2) | Approximately 3 years
  AUC0-t of revumenib and relevant metabolites (Phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Smith, M.D., Study Director — Syndax Pharmaceuticals
Locations (57):
- United States (22):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University Of California Care Medical Group - Norris Comprehensive Cancer Center And Hospital, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Florida Cancer Specialists and Research Institute, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa hospital, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
- Australia (5):
  - Peter MacCallum Cancer Centre (PMCC), Melbourne, Victoria
  - Royal Melbourne Hospital (RMH), Parkville, Victoria
  - Alfred Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal North Shore Hospital, Saint Leonards
- Canada (2):
  - University Health Network, Toronto
  - The Hospital for Sick Children, Toronto
- France (4):
  - Hospital Saint-Louis - APHP, Paris
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy-Gustave Roussy Cancer Center -DITEP, Villejuif
- Germany (7):
  - University Hospital Of Ulm, Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Essen (AoR), Essen
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitaetsmedizin Der Johannes, Gutenberg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - University of Leipzig, Leipzig
  - Klinikum Nuernberg Nord, Nuremberg
- Israel (6):
  - Rambam Health Care Campus (RHCC), Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center- Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (5):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Istituto Romagnolo Per Lo Studio dei tumori Dino Amadori, Meldola
  - IRCCS-Istituto Europeo di Oncologia, Milan
  - Universita Cattolica Fondazione Policlinico Agostino Gemelli, Roma
  - S Bortolo Hospital AULSS 8 Berica, Vicenza
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Princess Maxima Center for Pediatric Oncology, Utrecht, Netherlands
- Hospital Centro Comprensivo de Cancer UPR, San Juan, Puerto Rico
- Spain (3):
  - Institut Catala d'Oncologia (ICO) - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia MB, Wang B, Sheikh I, El Hajjar G, McCall D, Nunez C, Gibson A, Lorenzi PL, Issa GC, Cuglievan B, Abbas HA. High-throughput proteomic profiling to evaluate differentiation syndrome with menin inhibition. Mol Cell Proteomics. 2026 Jan 30:101522. doi: 10.1016/j.mcpro.2026.101522. Online ahead of print. PMID 41621809
- [Derived] Arellano ML, Thirman MJ, DiPersio JF, Heiblig M, Stein EM, Schuh AC, Zucenka A, de Botton S, Grove CS, Mannis GN, Papayannidis C, Perl AE, Issa GC, Aldoss I, Bajel A, Dickens DS, Kuhn MWM, Mantzaris I, Raffoux E, Traer E, Amitai I, Dohner H, Greco C, Kovacsovics T, McMahon CM, Montesinos P, Pigneux A, Shami PJ, Stone RM, Wolach O, Harpel JG, Chudnovsky Y, Yu L, Bagley RG, Smith AR, Blachly JS. Menin inhibition with revumenib for NPM1-mutated relapsed or refractory acute myeloid leukemia: the AUGMENT-101 study. Blood. 2025 Aug 28;146(9):1065-1077. doi: 10.1182/blood.2025028357. PMID 40332046
- [Derived] Issa GC, Aldoss I, Thirman MJ, DiPersio J, Arellano M, Blachly JS, Mannis GN, Perl A, Dickens DS, McMahon CM, Traer E, Zwaan CM, Grove CS, Stone R, Shami PJ, Mantzaris I, Greenwood M, Shukla N, Cuglievan B, Kovacsovics T, Gu Y, Bagley RG, Madigan K, Chudnovsky Y, Nguyen HV, McNeer N, Stein EM. Menin Inhibition With Revumenib for KMT2A-Rearranged Relapsed or Refractory Acute Leukemia (AUGMENT-101). J Clin Oncol. 2025 Jan;43(1):75-84. doi: 10.1200/JCO.24.00826. Epub 2024 Aug 9. PMID 39121437
- [Derived] Issa GC, Aldoss I, DiPersio J, Cuglievan B, Stone R, Arellano M, Thirman MJ, Patel MR, Dickens DS, Shenoy S, Shukla N, Kantarjian H, Armstrong SA, Perner F, Perry JA, Rosen G, Bagley RG, Meyers ML, Ordentlich P, Gu Y, Kumar V, Smith S, McGeehan GM, Stein EM. The menin inhibitor revumenib in KMT2A-rearranged or NPM1-mutant leukaemia. Nature. 2023 Mar;615(7954):920-924. doi: 10.1038/s41586-023-05812-3. Epub 2023 Mar 15. PMID 36922593
- [Derived] Sasca D, Guezguez B, Kuhn MWM. Next generation epigenetic modulators to target myeloid neoplasms. Curr Opin Hematol. 2021 Sep 1;28(5):356-363. doi: 10.1097/MOH.0000000000000673. PMID 34267079
- [Derived] Jimenez JA, Apfelbaum AA, Hawkins AG, Svoboda LK, Kumar A, Ruiz RO, Garcia AX, Haarer E, Nwosu ZC, Bradin J, Purohit T, Chen D, Cierpicki T, Grembecka J, Lyssiotis CA, Lawlor ER. EWS-FLI1 and Menin Converge to Regulate ATF4 Activity in Ewing Sarcoma. Mol Cancer Res. 2021 Jul;19(7):1182-1195. doi: 10.1158/1541-7786.MCR-20-0679. Epub 2021 Mar 19. PMID 33741715
- See also: Related Info — https://www.nature.com/articles/s41586-023-05812-3
- See also: Related Info — https://www.nature.com/articles/s41586-023-05755-9